CLINICAL TRIAL: NCT06036875
Title: CARE: Cancer Risk Perception and Women of Color
Status: Recruiting | Type: Observational
Sponsor: Mayo Clinic (Other)
Responsible Party: Sponsor
Other Study IDs: 22-012888; NCI-2023-04394 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 22-012888 (Other: Mayo Clinic Institutional Review Board)
Record Dates: First submitted 2023-09-07; First posted 2023-09-14 (Actual); Last update posted 2025-10-07 (Actual); Status verified 2025-10

CONDITIONS: Breast Carcinoma
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Health Services Research: Patients complete a survey and may participate in an interview on study.
  Interventions: Other: Non-Interventional Study

INTERVENTIONS:
Other: Non-Interventional Study — Non-interventional study

SUMMARY:
This study examines patient understanding of current and lifetime risk for breast cancer in women of color from diverse racial and ethnic backgrounds.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Examine the association between BC risk factors and BC risk perceptions among younger Black and Hispanic women and explore differences in associations by race and ethnicity (Black Hispanic, Black, Hispanic).

II. Explore how younger Black and Hispanic women conceptualize and formulate their risk for BC and to explore the relationship between risk perceptions and risk-reduction strategies.

OUTLINE: This is an observational study.

Patients complete a survey and may participate in an interview on study.

ELIGIBILITY:
Inclusion Criteria:

* Self-identify as female
* Between the ages of 18 and 50
* No medical history of breast cancer

Exclusion Criteria:

* Unable to understand or comprehend English or Spanish

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Self-identify as female
Study Population: Diverse women between 18 and 50 years of age
Sampling Method: Non-Probability Sample
Enrollment: 550 (Estimated)
Dates: Start 2023-03-25 (Actual); Primary Completion 2028-02-23 (Estimated); Study Completion 2028-02-23 (Estimated)

PRIMARY OUTCOMES:
Perception of risk | Baseline (at enrollment)
  Measured using a 0-100% response (percent lifetime risk) and a 5-point verbal scale ranging from 'very low' to 'very high' (ordinal lifetime risk). Participants will also be asked to assess their risk compared to women their age with the response options of 'much lower', 'about the same', and 'much higher' (comparative risk likelihood).

CONTACTS AND LOCATIONS:
Overall Officials: Jessica D. Austin, PhD, Principal Investigator — Mayo Clinic
Locations (3):
- United States (3):
  - Mayo Clinic in Arizona, Scottsdale, Arizona
  - University of Arizona, Tucson, Arizona
  - Mayo Clinic in Florida, Jacksonville, Florida

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials